CLINICAL TRIAL: NCT01761409
Title: Epidemiological Analysis on Endometrial Cancer.
Brief Title: Epidemiological Analysis on Endometrial Cancer in Guangdong Province of China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yet-Sen University Cancer Center (Other); First People's Hospital of Foshan (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Meizhou People's Hospital (Other); Jiangmen Central Hospital (Other); Guangdong Provincial People's Hospital (Other); Guangzhou Panyu Central Hospital (Other); First People's Hospital, Shunde China (Other); Yuebei People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaomao Li, Professor of Department of Gynecology, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: EC-2000-2010
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Endometrial cancer is one of the most common gynecological cancers, and the incidence increasing in the world. However, there isn't any large sample data of endometrial cancer reported in China. Thus Endometrial cancer project of Guangdong province conduct a large multicentre clinical investigation about endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer project of Guangdong province is mainly conducted by the Department of Gynecology of the Third Affiliated Hospital of Sun Yet-sen University, and other 62 major hospitals in Guangdong province participate in this project. In this large multicentre clinical investigation, the endometrial cancer database including more than 10,000 cases has been established. Further the investigators will demonstrate the epidemiological characteristics, etiology, risk factors, clinical treatment and prognosis of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients who was diagnosed with endometrial carcinoma from 2000 to 2010 in Guangdong province of China;
* patients with intact clinical and pathological information

Exclusion Criteria:

* not included in the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who was diagnosed with endometrial carcinoma from 2000 to 2010 in Guangdong province of China
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2000-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | five years

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital,Sun Yet-sen University, Guangzhou, Guangdong, China